CLINICAL TRIAL: NCT01800084
Title: Impact of Reconstruction Method (Adaptive Statistical Iterative Reconstruction, Filtered Back Projection) Used in Computed Tomography on Bone Single-Photon- Emission-Computed-Tomography/Computed-Tomography Image Quality
Brief Title: Impact of Reconstruction Method (ASIR, FBP) Used in CT on Bone SPECT/CT Image Quality
Acronym: AsirTest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2012/LS-01; 2013-A00070-45 (Other: RCB number)
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: SPECT-CT
Keywords: ASIR; image acquisition; FBP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing SPECT-CT (Experimental): The patients in this study are scheduled for a SPECT-CT at the Nîmes University Hospital as part of their normal care regimen.
  Intervention: Device: Asir Image Acquisition
  Interventions: Device: Asir Image Acquisition

INTERVENTIONS:
Device: Asir Image Acquisition — In addition to their normal image acquisition, a supplementary image acquisition lasting approximately 20 seconds (i.e. an ASIR image acquisition) will be carried out for each patient.

SUMMARY:
The main objective of this study is to demonstrate the non-inferiority of SPECT image quality (as measured by the signal / noise ratio) obtained by ASIR reconstruction of very-low-dose CT acquisitions versus the quality of those obtained by filtered back projection (FBP) of low-dose CT acquisitions.

The lower limit of non-inferiority is set to -1, the average SPECT signal / noise ratio TEMP expected is between 5 and 6.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. Demonstrate the non-inferiority of image quality (as assessed by a Likert scale) obtained by ASIR-reconstruction-SPECT versus FBP-reconstruction (the lower-limit of non-inferiority is set at -0.5); B. Verify the non-inferiority of image quality (as measured by the signal / noise ratio)of CT images obtained by ASIR-reconstruction versus FBP-reconstruction (the lower-limit of non-inferiority is set at -0.2); C. Verify the non-inferiority of image quality (as assessed by the Likert scale) of CT images obtained by ASIR-reconstruction versus FBP-reconstruction (the lower limit of non-inferiority is set at -0.5); D. Check that the irradiation dose received by the patient is lower for the acquisition of images reconstructed with ASIR than for the acquisition of images reconstructed with FBP.

E. Check the concordance of two evaluations of image quality (Likert scale) made by nuclear medicine physicians (blinded to each other).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* A SPECT-CT exam is scheduled for the patient
* The patient is able to withstand an extended position with the arms behind the head for 15 minutes (i.e. patient is able to undergo a SPECT-CT exam)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or any kind of guardianship
* The patient refuses to sign the consent
* The patient has a contra-indication for a treatment necessary for this study (patient is not able to withstand an extended position with the arms behind the head for 15 minutes)
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Emergency situations
* Presence of osteosynthesis material (or any other material that would generate an artifact during SPECT-CT) in the spine
* Patient behaviour hampers image acquisition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05-28 (Actual); Study Completion 2014-05-28 (Actual)

PRIMARY OUTCOMES:
Spect signal (kBq) | 2 hours after inclusion (during SPECT-CT scan)
  The Spect signal is measure on a 1 cm^3 zone of vertebrae L3.
Spect noise (kBq) | 2 hours after inclusion (during SPECT-CT scan)
  The spect noise is carried out on a 1 cm^3 zone of the aorta

SECONDARY OUTCOMES:
CT signal (HU) | 2 hours after inclusion (during SPECT-CT scan)
  measured on a 1 cm^3 zone of the aorta
CT noise (HU) | 2 hours after inclusion (during SPECT-CT scan)
  measured on a 1 cm^3 zone of the aorta
Ratio of CT signal / CT noise | 2 hours after inclusion (during SPECT-CT scan)
Spect image quality Likert scale ranging from 1 to 5, Evaluation n°1 | 2 hours after inclusion (during SPECT-CT scan)
CT image quality Likert scale ranging from 1 to 5, Evaluation n°2 | 2 hours after inclusion (during SPECT-CT scan)
Radiation dose (mSv) | 2 hours after inclusion (during SPECT-CT scan)
Spect image quality Likert scale ranging from 1 to 5, Evaluation n°2 | 2 hours after inclusion (during SPECT-CT scan)
CT image quality Likert scale ranging from 1 to 5, Evaluation n°1 | 2 hours after inclusion (during SPECT-CT scan)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Sibille, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France

REFERENCES:
- [Result] Sibille L, Chambert B, Alonso S, Barrau C, D'Estanque E, Al Tabaa Y, Collombier L, Demattei C, Kotzki PO, Boudousq V. Impact of the Adaptive Statistical Iterative Reconstruction Technique on Radiation Dose and Image Quality in Bone SPECT/CT. J Nucl Med. 2016 Jul;57(7):1091-5. doi: 10.2967/jnumed.115.164772. Epub 2016 Mar 24. PMID 27013695